CLINICAL TRIAL: NCT04750889
Title: RFID Trial: Localization of Non-palpable Breast Lesions Using Radiofrequency Identification Tags or Wire
Brief Title: Breast Localization: RFID Tags vs Wire Localization
Acronym: RFID
Status: Completed | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Other Study IDs: RFID
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Neoplasm Female
Keywords: Non palpable breast cancer; RFID tags; Observational study; Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RFID tags localization
  Interventions: Device: RFID tags
- Wire localization
  Interventions: Device: Wire localization

INTERVENTIONS:
Device: RFID tags — Installation of the RFID tag device wire localization)
  Groups: RFID tags localization
Device: Wire localization — Installation of the wire localization device
  Groups: Wire localization

SUMMARY:
The RFID trial focuses on breast localization in patients with non-palpable breast cancers. It aims to demonstrate the improvement in patient comfort when using the Radio Frequency Identification (RFID) tag and LOCalizer™ device compared to the gold standard device.

DETAILED DESCRIPTION:
It is an observational, prospective, single-center, 2-arm (RFID group vs. standard gold), non-randomized and category 3 comparative study. The RFID trial focuses on breast localization in patients with non-palpable breast cancers. These patients will benefit from a mastology consultation: consent will then be acquired. The RFID tag or the gold standard localization will be put in place during this consultation (one day before surgery).

Patients will fill in their questionnaire in two steps:

* during the installation of the device (RFID tag or wire localization) to evaluate the patient's pain,
* then at the 1-month post-operative consultation to assess pain in the interval until surgery Radiologists and surgeons will fill out the questionnaire dedicated to them after each procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older,
* Requiring conservative surgical management for a breast lesion -infra-clinical (fibroadenomas, papillomas, atypical lesions, neoplasia), whose histology will have been proven beforehand by anatomopathology.
* Patients referred to mastology for preoperative identification by the surgeons
* Able to give informed consent to participate in the research.
* Affiliation to a Social Security regime

Exclusion Criteria:

* Multiple breast lesions
* Patients with breast neoplasia during pregnancy.
* Person deprived of liberty or under guardianship or incapable of giving consent
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age or older patients requiring conservative surgical management for a breast lesion infra-clinical (fibroadenomas, papillomas, atypical lesions, neoplasia), whose histology will have been proven beforehand by anatomopathology
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of the patients satisfaction | 1 years and 1 month
  The value of the satisfaction score of the patient questionnaire from 0 (worst statisfaction) to 10 (better statisfaction)

SECONDARY OUTCOMES:
Satisfaction of surgeons and radiologists assessed by a questionnaire | 1 years and 1 month
  overall score values from the surgeon and radiologist questionnaires
Evaluation of the quality of the RFID tag device by analizing surgery data | 1 years and 1 month
  the occurrence or not of a migration of the RFID tag, histological data, the invasion of the margins and the rate of reoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pete R, Pinard C, Sirodot F, Molnar I, Dressaire M, Ginzac A, Abrial C, Durando X, Tekath M. Patient satisfaction with radio-frequency identification (RFID) tag localization compared with wire localization for nonpalpable breast lesions: the RFID trial. BMC Cancer. 2025 Jan 22;25(1):123. doi: 10.1186/s12885-025-13453-0. PMID 39844175
- [Derived] Veyssiere H, Dressaire M, Pete R, Pinard C, Molnar I, Abrial C, Ginzac A, Durando X, Tekath M. RFID trial: localization of non-palpable breast lesions using radiofrequency identification tags or wire. BMC Cancer. 2023 Jul 20;23(1):679. doi: 10.1186/s12885-023-11190-w. PMID 37468859